CLINICAL TRIAL: NCT01362335
Title: Electronic Registration of Noninvasively Acquired Hemodynamic Parameters Using Nexfin®-Monitoring System
Brief Title: Nexfin®-Monitoring System
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: Nex-001
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients, that are having a routine surgical procedure.

SUMMARY:
In many surgical procedures, anaesthesiological care is provided according to the best scientific and clinical information available. However, since hemodynamic monitoring until recently did not allow for beat-to-beat information of the haemodynamical changes, many fast-changing events may have been unnoticed or have not been investigated as precisely as is possible today. Moreover, in several surgical procedures - like eye surgery - the invasiveness of the classical haemodynamical monitoring devices was of such a degree that until now, in these circumstances these vital parameters were not investigated yet.

Therefore, the availability of this new device, which allows for noninvasive beat-to-beat assessment of these haemodynamical parameters gives a unique opportunity to investigate our anaesthesiological management and to elucidate whether improvements are desirable and possible.

The Nexfin monitor consists of a cuff-micromanometer that is located around the third finger. It simultaneously uses continuous pressure readings and light-absorption spectrometry to determine valuable haemodynamical information. Data is recorded and available for subsequent offline analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are accepted for surgery

Exclusion Criteria:

* Patients unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, that are having a routine surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
haemodynamical changes after several surgical and anaesthesiological interventions. | 30 minutes - 2 hours
  Beat-to-beat determination of stroke volume, cardiac output, blood pressure and systemic resistance measurement

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Vos JJ, Poterman M, Mooyaart EA, Weening M, Struys MM, Scheeren TW, Kalmar AF. Comparison of continuous non-invasive finger arterial pressure monitoring with conventional intermittent automated arm arterial pressure measurement in patients under general anaesthesia. Br J Anaesth. 2014 Jul;113(1):67-74. doi: 10.1093/bja/aeu091. Epub 2014 Apr 15. PMID 24740992